CLINICAL TRIAL: NCT02981823
Title: Effect of Periprosthetic Fracture on Hip Function After Femoral Neck-preserving Total Hip Arthroplasty: a Prospective, Single-center, Self-controlled Trial With 2-year Follow-up
Brief Title: Effect of Periprosthetic Fracture on Hip Function After Femoral Neck-preserving Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HebeiMUTH_QD_001
Record Dates: First submitted 2016-11-24; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hip replacement (Experimental): The patients undergo total hip replacement with the collum femoris preserving stem suffered from periprosthetic fractures.
  Interventions: Procedure: hip replacement

INTERVENTIONS:
Procedure: hip replacement — The patients undergo hip replacement with the collum femoris preserving stem suffered from periprosthetic fractures.

SUMMARY:
To provide information on reducing the incidence of periprosthetic fractures during hip replacement with the CFP prosthetic stem by analyzing the risk factors for periprosthetic fractures and their effects on hip functional recovery.

DETAILED DESCRIPTION:
History and current related studies Periprosthetic fractures are one of the challenges for orthopedic surgeons that are more likely to appear during hip replacement with a cementless prosthesis. Hip replacement with a collum femoris preserving (CFP) prosthetic stem allows the preservation of the femoral neck and preserves bone tissues as much as possible for prosthetic revision in the future. However, the occurrence of periprosthetic fractures will result in a failure surgery. Existing evidence has shown that although hip replacement with the CFP prosthetic stem can reduce complications and pain, periprosthetic fractures that are more likely to occur during the surgery badly impact functional recovery in patients.

Adverse events Adverse events which occurred during the follow-up, including hip pain, prosthetic loosening, spinal cord and nerve injuries, soft tissue infection and poor prosthetic position, were recorded.

If severe adverse events occurred during the follow-up, their details including the date of occurrence, type of adverse events and measures taken were recorded and reported to the principal investigator and the institutional review board within 24 hours.

Data collection, management, analysis, and open access Data collection Clinical data, including demographic data, disease diagnosis, accompanying diseases, allergic history (drug allergy) and adverse events, were collected and summarized using standardized case report forms. These data were processed using Epidata software and electronically input using double entry system.

Data management After database confirmation, only the project manager was able to access the database. The locked data were unable to be altered and were preserved by the Third Hospital of Hebei Medical University.

Data analysis All data were statistically analyzed by professional statisticians who were responsible for completing an outcome analysis report that was submitted to the project manager. An independent data monitoring committee was responsible for data monitoring and management throughout the entire trial to ensure scientific accuracy, stringency, authenticity, and integrity.

Statistical analysis All data were statistically analyzed by statisticians using SPSS 21.0 software in line with the intention-to-treat principle. Normally distributed measurement data were expressed as means, standard deviations, minimums, and maximums, while non-normally distributed data were expressed as lower quartiles, medians, and upper quartiles.

Wilcoxon matched paired test was used for comparative analysis of Harris hip scores and imaging parameters as determined before and 6, 12, 24 months after operation. Then, a multivariate logistic regression analysis was used to calculate the regression coefficient, OR, 95% CI with the Harris scale as the dependent variable for each imaging parameter which had significant difference. The statistical significance level was α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and staging criteria in line with the Expert consensus on diagnosis and treatment of adult femoral head necrosis
* Femoral head necrosis of Association Research Circulation Osseous (ARCO) stages III-IV
* Unilateral femoral head necrosis
* Age < 50 years
* Both genders

Exclusion Criteria:

* Advanced osteoarthritis
* Secondary osteoarthritis due to acetabular dysplasia
* Ankylosing spondylitis involving the hip joint
* Rheumatoid arthritis
* Inflammatory inflammation of the hip joint
* Tumor lesions in the hip joint
* Unable or refusal to sign the informed consent

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Harris hip scores | Changes of baseline and 6 months after operation
  To evaluate the recovery of hip joint function. Harris hip scores have a range of 0-100 points: excellent ≥ 90 points, good 80-89 points, fair 70-79 points, and poor <70 points. The higher score indicates the better function of the hip.

SECONDARY OUTCOMES:
X-ray image | Changes of baseline and month 6, month 12, month 24 after operation
  To observe anteroposterior and frog-leg lateral X-ray films of the hip as well as full-length X-ray films of the bilateral lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Di Qin, Ph.D, Principal Investigator — Hebei Medical University Third Hospital

IPD SHARING:
Plan to Share IPD: No